CLINICAL TRIAL: NCT04962451
Title: Efficacy and Safety of Ticagrelor Combined With ASA Versus ASA Alone in Preventing Stroke and Death in Patients With Acute Ischemic Stroke or Transient Ischemic Attack: a Randomized, Double-blind, Placebo-controlled, International Multicenter Phase III Clinical Study
Brief Title: Comparison of the Efficacy of Ticagrelor Combined With ASA to ASA Alone in Patients With Stroke
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D2017121
Record Dates: First submitted 2021-06-27; First posted 2021-07-15 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-06

CONDITIONS: Cerebrovascular Accident; Cerebrovascular Accident, Acute
MeSH Terms: conditions — Stroke | interventions — Ticagrelor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Drug: ticagrelor + ASA
- Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo+ASA

INTERVENTIONS:
Drug: ticagrelor + ASA — On day 1, ticagrelor loading dose (2 tablets, ticagrelor 90mg) was given, followed by ticagrelor 90mg, twice daily Basic treatment: the first day received ASA loading dose, 300-325mg, and the server received ASA 75-100mg, once a day
  Arms: Intervention group
Drug: Placebo+ASA — Placebo loading dose on day 1 (2 tablets, matched with ticagrelor 90mg), followed by placebo twice daily (matched with ticagrelor 90mg) Basic treatment: the first day received ASA loading dose, 300-325mg, and the server received ASA 75-100mg, once a day
  Arms: Placebo group

SUMMARY:
Cerebrovascular disease is the main cause of death and severe long-term disability worldwide. Antiplatelet drugs are the main drugs for ischemic stroke and TIA. Cyclooxygenase inhibitor acetylsalicylic acid (ASA) has always been the most widely studied antiplatelet therapy. The studies of acrates of aliscon body evaluated the efficacy and safety of ticagrelor monotherapy in preventing major vascular events in patients with AIS or TIA. The results showed that the number of patients with endpoint events in ticagrelor group was less than that in ASA group, However, it has not been proved that ticagrelor monotherapy is better than ASA. The purpose of this study is to prove that ticagrelor is better than ASA.

DETAILED DESCRIPTION:
Cerebrovascular disease is the main cause of death and severe long-term disability worldwide. Antiplatelet drugs are the main drugs for ischemic stroke and TIA. Cyclooxygenase inhibitor acetylsalicylic acid (ASA) has always been the most widely studied antiplatelet therapy. The studies of acrates of aliscon body evaluated the efficacy and safety of ticagrelor monotherapy in preventing major vascular events in patients with AIS or TIA. The results showed that the number of patients with endpoint events in ticagrelor group was less than that in ASA group, However, it has not been proved that ticagrelor monotherapy is better than ASA. The purpose of this study is to prove that ticagrelor is better than ASA. The study will be designed as a randomized, double-blind, placebo-controlled, parallel grouping study and conducted in multiple centers to ensure the representation of multiple countries, races and races, so as to ensure that the results of the study can be widely applied.

ELIGIBILITY:
Inclusion Criteria:

1. Over 40 years old
2. Acute ischemic attack
3. Symptoms occurred within 24 hours after randomization

Exclusion Criteria:

1. Dual antiplatelet therapy with ASA and P2Y12 inhibitors is needed
2. Antiplatelet agents other than ASA
3. Anticoagulant therapy
4. Have any atrial fibrillation / flutter
5. Renal failure requiring dialysis
6. During pregnancy or lactation

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13000 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events | At day 7 after participants included into the research
  The event that patients have stroke or die
Occurrence of adverse events | At day 30 after participants included into the research
  The event that patients have stroke or die
Occurrence of adverse events | At day 60 after participants included into the research
  The event that patients have stroke or die

SECONDARY OUTCOMES:
Tool assessment result | At day 60 after participants included into the research
  Score of Modified Rankin Scale

CONTACTS AND LOCATIONS:
Overall Officials: Xiaogang Li, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No